CLINICAL TRIAL: NCT01655563
Title: A Pharmacogenetic Trial of Tacrolimus Dosing After Pediatric Transplantation
Brief Title: Pharmacogenetic Trial of Tacrolimus After Pediatric Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Seema Mital, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000026524
Record Dates: First submitted 2012-07-27; First posted 2012-08-02 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Heart Transplantation; Liver Transplantation; Kidney Transplantation
Keywords: Transplant; Pediatrics; Tacrolimus; Prograf
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Dosing Arm (Active Comparator): Patients in the standard arm will receive standard starting dose of tacrolimus that is clinically used i.e. 0.1 mg/kg/dose twice a day.
  Interventions: Drug: Tacrolimus
- Pharmacogenetic Arm (Experimental): Patients in the pharmacogenetic arm will receive a starting dose that is assigned based on age and CYP3A5 expressor status. Patients that are CYP3A5 expressors will receive the higher end of the dose range compared to non-expressors. All doses recommended represent clinically acceptable and safe dose ranges used at our institution.
  CYP3A5 non-expressor starting dose:
  Greater than 6 years of age - 0.075 mg/kg/dose q12 hours; Less than or equal to 6 years of age - 0.1 mg/kg/dose q12 hours
  CYP3A5 expressor starting dose:
  Greater than 6 years of age - 0.15 mg/kg/dose q12 hours; Less than or equal to 6 years of age - 0.2 mg/kg/dose q12 hours
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus, a calcineurin inhibitor, is the commonest immunosuppressive agent used for maintenance immunosuppression after solid organ transplantation. The mechanism of action involves binding to an intracellular protein, FKBP-12. A complex of tacrolimus-FKBP-12, calcium, calmodulin and calcineurin is then formed and the phosphatase activity of calcineurin is inhibited. This prevents the generation of nuclear factor of activated T-cells, a nuclear component, resulting in inhibition of transcription of lymphokines (interleukin-2, γ-interferon). The net result is the inhibition of T-lymphocyte activation.Tacrolimus is metabolized primarily by the CYP3A enzymes in the liver particularly the CYP3A5.
  Other Names: Prograf

SUMMARY:
Tacrolimus is a standard and widely used maintenance immunosuppressive agent after solid organ transplantation.The purpose of this trial is to determine if dosing of tacrolimus through genetics will help in early attainment and maintenance of the correct dosage level in the early post-transplant period. This pilot dose-finding trial will help to determine a dosing strategy guided by genotypes and age for solid organ transplant recipients that will be further validated through a multi-centre trial as an immediate next step. The study hypothesizes that dosage levels determined through age and genotype will be attained faster and more accurately than the standard dosing procedures in the 14-days after the transplant. Further, this study hypothesizes that a genotype and age dosing strategy will cause a faster recovery (tested through the kidneys' ability to clear creatine from the blood) and result in lower frequencies of adverse effects and rejection of the transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years old
* Assessed and/or listed for heart, kidney, liver transplantation
* Planned oral or enteral maintenance immunosuppression with tacrolimus post transplant
* Informed consent of legal guardian

Exclusion Criteria:

* Contra-indications to oral or enteral tacrolimus
* Co-morbidities that preclude standard dosing e.g. significant renal or hepatic insufficiency
* Participation in other investigational drug trials within 30 days of study initiation

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Mital, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Min S, Papaz T, Lafreniere-Roula M, Nalli N, Grasemann H, Schwartz SM, Kamath BM, Ng V, Parekh RS, Manlhiot C, Mital S. A randomized clinical trial of age and genotype-guided tacrolimus dosing after pediatric solid organ transplantation. Pediatr Transplant. 2018 Nov;22(7):e13285. doi: 10.1111/petr.13285. Epub 2018 Sep 3. PMID 30178515

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 participants were excluded after enrollment due to the following reasons: 8 developed ineligibility criteria for randomization, 2 withdrew, 4 were delisted for transplant, 4 died and 4 had still not received a transplant.
Period: Overall Study
Arm/Group | Standard Dosing Arm | Pharmacogenetic Arm
Started | 18 | 35
Completed | 18 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 53 patients were randomized, 35 to the pharmacogenetic arm (6 CYP3A5 expressors, 29 CYP3A5 non-expressors) and 18 to the standard dosing arm.
Groups:
- Pharmacogenetic Arm: Patients in the pharmacogenetic arm will receive a starting dose that is assigned based on age and CYP3A5 expressor status. Patients that are CYP3A5 expressors will receive the higher end of the dose range compared to non-expressors as described in Table 1. All doses recommended in Table 1 represent clinically acceptable and safe dose ranges used at our institution. This proposed pharmacogenetic dosing algorithm is derived from a validated algorithm published in pediatric renal transplant patients.
- Total: Total of all reporting groups
Arm/Group | Standard Dosing Arm | Pharmacogenetic Arm | Total
Number analyzed (Participants) | 18 | 35 | 53
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age at transplant was collected
  years | 1.3 [0.8 to 5.9] | 2.8 [0.7 to 13.5] | 2.1 [0.75 to 8.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 5 | 19 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 26 | 38
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 35 | 53

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Therapeutic Tacrolimus Drug Concentrations
Description: The primary outcome (efficacy) was time to achieve therapeutic tacrolimus trough concentrations
Time Frame: From Baseline to 30 days post-dose
Population: The overall number of participants analyzed was 53. A total of 7 patients (4 from genotype-guided dosing arm and 3 from standard dosing arm) began but did not complete 36- 48 hours of study dosing and were analyzed in their original assigned groups in an intention-to- treat model.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Standard Dosing Arm | Pharmacogenetic Arm
Number analyzed (Participants) | 18 | 35
Days | 4.7 [3.5 to 8.6] | 3.4 [2.5 to 6.6]

2. Primary Outcome: Time to Maintain Stable Therapeutic Trough Concentrations
Description: Defined as two consecutive concentrations at least 48 hours apart in the therapeutic range without any changes in tacrolimus dose
Time Frame: From Baseline to 30 days post-dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Dosing Arm | Pharmacogenetic Arm
Number analyzed (Participants) | 18 | 35
days | NA [NA to NA] — Median time could not be generated for the standard dosing arm because <50% participants achieved stable therapeutic concentration during study follow-up leading to an insufficient number of participants with events. | 18 [14 to 27]

3. Secondary Outcome: Clinical Adverse Events
Description: The effect of pharmacogenetic dosing of tacrolimus for 48 hours on the frequency clinical adverse effects over 30±3 days.
Time Frame: Over 30 days, +/- 3 days
Population: as for outcome 1
Measure: Number; unit: adverse events
Arm/Group | Standard Dosing Arm | Pharmacogenetic Arm
Number analyzed (Participants) | 18 | 35
adverse events | 71 | 121

ADVERSE EVENTS:
Time Frame: Baseline to 30 days post transplant
Description: AEs were classified by intensity, severity, relationship to investigational agent, expectedness of the event, treatment or action taken, and clinical outcome. All serious, unexpected adverse drug reactions to the study medication were reported to Health Canada within 15 calendar days or for death or life-threatening events, within 7 calendar days. A copy of any serious, unexpected adverse drug reaction reports was sent to the Data and Safety Monitoring Committee.
Arm/Group | Standard Dosing Arm | Pharmacogenetic Arm
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/18 | 4/35
Other Adverse Events (participants affected / at risk) | 18/18 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dosing Arm (N=18) | Pharmacogenetic Arm (N=35)
Pericardial hematoma (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased LFTs (Hepatobiliary disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Reactive airway disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
IVC thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dosing Arm (N=18) | Pharmacogenetic Arm (N=35)
Hypertension (Vascular disorders) | 10 (11) | 15 (15)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Arrthythmia (Cardiac disorders) | 2 (2) | 4 (4)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 4 (4)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Viremia (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 6 (6)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 3 (3)
Allergic reaction (Immune system disorders) | 4 (4) | 1 (1)
Rejection/ suspected rejection (Immune system disorders) | 4 (4) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Blood tacrolimus level increased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase and/or aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 4 (4)
Edema face/limbs/ trunk (General disorders) | 1 (1) | 4 (4)
pain in extremity (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The current trial was a pilot trial for feasibility, safety and preliminary efficacy. It was not powered to study confounding influence of other recipient factors and of donor genotype on outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes